CLINICAL TRIAL: NCT00762177
Title: Investigate Oral Bacteria in Adult Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRO-0108-BACT-PS-NJ
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-02

CONDITIONS: Oral Bacteria
MeSH Terms: interventions — Fluorides; Triclosan; hydrated silica gel-based toothpaste; Tin Fluorides

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A -Control (Placebo Comparator): fluoride toothpaste
  Interventions: Drug: Fluoride
- B Experimental toothpaste (Experimental): Stannous fluoride toothpaste
  Interventions: Drug: Stannous Fluoride
- C- positive control (Active Comparator): fluoride/triclosan/copolymer toothpaste
  Interventions: Drug: Fluoride, Triclosan

INTERVENTIONS:
Drug: Fluoride — Brush twice a day for 14 days
  Other Names: Crest Anti-Cavity toothpaste
  Arms: A -Control
Drug: Fluoride, Triclosan — Brush twice daily for 14 days
  Other Names: Total toothpaste
  Arms: C- positive control
Drug: Stannous Fluoride — Brush twice daily for 14 days
  Arms: B Experimental toothpaste

SUMMARY:
To compare the antimicrobial efficacy of three dentifrices on oral bacteria

ELIGIBILITY:
Inclusion Criteria:

* Males and females in good general health aged 18 to 70 years.
* A willingness to read, understand, and sign the Informed Consent Form after the nature of the study has been fully explained to them. Subject should demonstrate a willingness to comply with all study procedures and sampling schedules.
* A minimum of 20 natural teeth with facial and lingual scorable surfaces.
* Adequate oral hygiene and no signs of oral neglect.
* Good periodontal health. Enrolled subjects will have periodontal pockets no greater than 5 mm.
* Gingival and plaque indices will also be measured during the first visit. Subjects with gingival index greater than or equal to 1.5 (Lobene Index) and plaque index greater than or equal to 1.5 (Turesky modification of Quigley-Hein Index) will be enrolled.

Exclusion Criteria:

* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses. Allergy to personal care/consumer products or their ingredients. Previous known allergy to dental materials, particularly to acrylic-like materials used to fabricate the stent device (this is a highly unlikely occurrence).
* Teeth that are grossly carious, fully crowned or extensively restored on facial and/or lingual surfaces, orthodontically banded, abutments, or third molars
* Difficulty having dental impressions taken such as excessive gagging.
* History of diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases, e.g. heart disease or AIDS.
* History of rheumatic fever, heart murmur, mitral valve prolapse or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
* Subjects on antibiotic, antiinflammatory or anticoagulant therapy during the month preceding the baseline exam.
* Significant oral soft tissue pathology, systemically related gingival enlargement, severe gingivitis (based on a visual examinations).
* History of active severe periodontal disease with bleeding gums and loose teeth.
* Gross dental caries, severe generalized cervical abrasion and/or enamel abrasion, large fractured or temporary restorations (based on visual examinations).will not be included in the tooth count.
* Fixed or removable orthodontic appliance or removable partial dentures.
* Participation in a dental plaque/gingivitis clinical study involving oral care products, within the last 30 days. History of dental prophylaxis or treatments in the past month.
* Self reported pregnancy or lactation.
* History or current use of objects to pierce the lips or tongue.
* Subjects known to be an alcoholic, or a recovering alcoholic.
* History or current use of recreational drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fine, DDS, Principal Investigator
Locations (1):
- Department of Oral Biology, Newark, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited by the PI at the clinical site
Pre-assignment Details: Subjects were screened for medical and oral health criteria and then entered a 1 week washout.
Groups:
- Placebo 1st, Active Comparator 2nd and Experimental 3rd: Participants brushed their teeth with the placebo control (fluoride toothpaste only)during the first intervention then brushed with active comparator(fluoride/triclosan/copolymer toothpaste) during the second intervention and experimental product (stannous fluoride toothpaste) during as the last intervention.
- Active Comparator 1st, Experimental 2nd, Placebo 3rd: Participants brushed their teeth with the Active Comparator (fluoride/triclosan/copolymer toothpaste)during the first intervention, then brushed with experimental product (stannous fluoride toothpaste) during the second intervention, and brushed with the placebo control (fluoride toothpaste only)as the last intervention.
- Experimental 1st, Placebo 2nd, Active Comparator 3rd: Participants brushed their teeth with the experimental product (stannous fluoride toothpaste) during the first intervention, then brushed with the placebo control (fluoride toothpaste only) during the second intervention and Active Comparator(fluoride/triclosan/copolymer toothpaste)as the last intervention.
Period: 1st Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental 3rd | Active Comparator 1st, Experimental 2nd, Placebo 3rd | Experimental 1st, Placebo 2nd, Active Comparator 3rd
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Washout After 1st Treatment
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental 3rd | Active Comparator 1st, Experimental 2nd, Placebo 3rd | Experimental 1st, Placebo 2nd, Active Comparator 3rd
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: 2nd Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental 3rd | Active Comparator 1st, Experimental 2nd, Placebo 3rd | Experimental 1st, Placebo 2nd, Active Comparator 3rd
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Washout After 2nd Treatment
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental 3rd | Active Comparator 1st, Experimental 2nd, Placebo 3rd | Experimental 1st, Placebo 2nd, Active Comparator 3rd
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: 3rd Treatment Period
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental 3rd | Active Comparator 1st, Experimental 2nd, Placebo 3rd | Experimental 1st, Placebo 2nd, Active Comparator 3rd
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo 1st, Active Comparator 2nd and Experimental 3rd | Active Comparator 1st, Experimental 2nd, Placebo 3rd | Experimental 1st, Placebo 2nd, Active Comparator 3rd | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.87 (10.72) | 40.12 (9.38) | 36.5 (7.46) | 38.83 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 4 | 16
  Male | 1 | 3 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Species in Plaque(Actinomyces)
Description: After 14 days of study product use, dental plaque was scraped from the subject's teeth. The plaque was placed in sterile phosphate buffered saline(PBS) and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on CFAT Agar
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Groups:
- Placebo Toothpaste: Participants brushed their teeth with the placebo control (fluoride toothpaste only).
- Active Comparator: Participants brushed their teeth with the Active Comparator(fluoride/triclosan/copolymer toothpaste).
- Experimental: Participants brushed their teeth with the experimental product (stannous fluoride toothpaste).
Arm/Group | Placebo Toothpaste | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | 0.023 (0.0478) | 0.3881 (0.322) | 0.0538 (0.0247)
Statistical Analysis 1: Comparison: Placebo Toothpaste vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Antimicrobial Species in Saliva(Actinomyces)
Description: Saliva was collected, after 14 days of product use, by drooling into a tube and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in sterile phosphate buffered saline(PBS) and plated using a spiral systems autoplate 4000 spiral plater on CFAT Agar
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Groups:
- Placebo: Participants brushed their teeth with the placebo control (fluoride toothpaste only)
- Active Comparator: Participants brushed their teeth with the Active Comparator (fluoride/triclosan/copolymer toothpaste).
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | 0.016 (0.0236) | 0.3209 (0.0301) | 0.1116 (0.0272)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

3. Primary Outcome: Antimicrobial Species on the Tongue(Actinomycetes)
Description: After 14 days of study product use, the tongue was scraped 5 times with the edge of a tongue depressor. The sample is vortexed in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on CFAT Agar
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0132 (0.0229) | 0.2612 (0.0402) | -0.0536 (0.0262)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

4. Primary Outcome: Antimicrobial Species on the Cheek(Actinomyces)
Description: After 14 days of study product use, the inside of the cheek was scraped with a swab and place in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on CFAT Agar
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | 0.0099 (0.027) | 0.2949 (0.0327) | -0.1875 (0.0354)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

5. Primary Outcome: Antimicrobial Species in Plaque(Total Anaerobic)
Description: After 14 days of study product use, dental plaque scraped from teeth, placed in sterile phosphate buffered saline(PBS) and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on ETSA Agar
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0629 (0.0475) | 0.312 (0.0404) | 0.0762 (0.0547)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

6. Primary Outcome: Antimicrobial Species in Saliva(Total Anaerobic)
Description: After 14 days of study product use, saliva was collected by drooling into a tube and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in sterile phosphate buffered saline(PBS) and plated using a spiral systems autoplate 4000 spiral plater on ETSA Agar
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0247 (0.0266) | 0.1505 (0.0298) | 0.05 (0.0331)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

7. Primary Outcome: Antimicrobial Species in Tongue(Total Anaerobic)
Description: After 14 days of study product use, the tongue was scraped 5 times with the edge of a tongue depressor. The sample is vortexed in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on ETSA Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0445 (0.0508) | 0.2691 (0.0403) | 0.0926 (0.0334)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

8. Primary Outcome: Antimicrobial Species on the Cheek(Total Anaerobic)
Description: After 14 day of study product use, the inside of the cheek was scraped with a swab and place in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on ETSA Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0551 (0.0259) | 0.2009 (0.038) | -0.0531 (0.0346)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; the tongue will be scrapped 5 times with the edge of a tongue depressor. The depressor is vortex in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on CFAT Agar; Test type: Superiority or Other; p = 0.05, ANCOVA

9. Primary Outcome: Antimicrobial Species in Plaque(Fusobacteria)
Description: After 14 days of study product use, dental plaque scraped from teeth, placed in sterile phosphate buffered saline(PBS) and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on CVE Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.2973 (0.0503) | 0.2703 (0.0431) | -0.0095 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

10. Primary Outcome: Antimicrobial Species in Saliva(Fusobacteria)
Description: After 14 days of study product use, saliva was collected by drooling into a tube and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in sterile phosphate buffered saline(PBS) and plated using a spiral systems autoplate 4000 spiral plater on CVE Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0096 (0.0265) | 0.194 (0.0356) | 0.0539 (0.0311)
Statistical Analysis 1: Comparison: Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

11. Primary Outcome: Antimicrobial Species in Tongue(Fusobacteria)
Description: After 14 days of study product use, the tongue was scraped 5 times with the edge of a tongue depressor. The sample is vortexed in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on CVE Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0742 (0.0416) | 0.377 (0.0495) | 0.1668 (0.048)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

12. Primary Outcome: Antimicrobial Species on the Cheek(Fusobacteria)
Description: After 14 days of study product use, the inside of the cheek was scraped with a swab and place in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on CVE Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0319 (0.0458) | 0.1887 (0.0251) | 0.111 (0.0265)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

13. Primary Outcome: Antimicrobial Species in Plaque(Oral Streptococci)
Description: After 14 days of study product use, dental plaque scraped from teeth, placed in sterile phosphate buffered saline(PBS) and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on Mitis Salivarius Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0848 (0.0417) | 0.2593 (0.043) | -0.0096 (0.0358)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

14. Primary Outcome: Antimicrobial Species in Saliva(Oral Streptococci)
Description: After 14 days of study product use, saliva was collected by drooling into a tube and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in sterile phosphate buffered saline(PBS) and plated using a spiral systems autoplate 4000 spiral plater on Mitis Salivarius Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0436 (0.0307) | 0.1445 (0.0305) | 0.087 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

15. Primary Outcome: Antimicrobial Species in Tongue(Oral Streptococci)
Description: After 14 days of study product use, the tongue was scraped 5 times with the edge of a tongue depressor. The sample is vortexed in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on Mitis Salivarius Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.1284 (0.0537) | 0.2233 (0.0355) | 0.0525 (0.0358)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

16. Primary Outcome: Antimicrobial Species on the Cheek(Oral Streptococci)
Description: After 14 days of study product use, the inside of the cheek was scraped with a swab and place in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on Mitis Salivarius Agar
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | 0.0126 (0.0326) | 0.2088 (0.0388) | -0.0251 (0.0309)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

17. Primary Outcome: Antimicrobial Species in Plaque(Sulfur Bacteria)
Description: After 14 days of study product use, dental plaque scraped from teeth, placed in sterile phosphate buffered saline(PBS) and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on OHO Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | 0.0174 (0.0625) | 0.3083 (0.0424) | -0.0416 (0.057)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

18. Primary Outcome: Antimicrobial Species in Saliva(Sulfur Bacteria)
Description: After 14 days of study product use, saliva was collected by drooling into a tube and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in sterile phosphate buffered saline(PBS) and plated using a spiral systems autoplate 4000 spiral plater on OHO Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.1213 (0.0494) | 0.1556 (0.0375) | -0.603 (0.0315)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

19. Primary Outcome: Antimicrobial Species in Tongue(Sulfur Bacteria)
Description: After 14 days of study product use, the tongue was scraped 5 times with the edge of a tongue depressor. The sample is vortexed in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on OHO Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.083 (0.0564) | 0.2065 (0.0474) | -0.0248 (0.0511)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

20. Primary Outcome: Antimicrobial Species on the Cheek(Sulfur Bacteria)
Description: After 14 days of study product use, the inside of the cheek was scraped with a swab and place in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on OHO Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.1788 (0.0362) | 0.2036 (0.0581) | -0.0815 (0.0373)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

21. Primary Outcome: Antimicrobial Species in Plaque(Veillonella)
Description: After 14 days of study product use, dental plaque scraped from teeth, placed in sterile phosphate buffered saline(PBS) and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on Veillonella Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | 0.0007 (0.0478) | 0.3658 (0.0322) | 0.0316 (0.0247)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

22. Primary Outcome: Antimicrobial Species in Saliva(Veillonella)
Description: After 14 days of study product use, saliva was collected by drooling into a tube and sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in sterile phosphate buffered saline(PBS) and plated using a spiral systems autoplate 4000 spiral plater on veillonella Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | 0.0167 (0.0213) | 0.3062 (0.0305) | 0.0901 (0.0261)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

23. Primary Outcome: Antimicrobial Species in Tongue(Veillonella)
Description: After 14 days of study product use, the tongue was scraped 5 times with the edge of a tongue depressor. The sample is vortexed in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on Veillonella Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.002 (0.0229) | 0.2724 (0.0402) | -0.0424 (0.0262)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

24. Primary Outcome: Antimicrobial Species on the Cheek(Veillonella)
Description: After 14 days of study product use, the inside of the cheek was scraped with a swab and place in sterile phosphate buffered saline(PBS) and the sample is then sonicated using a Branson 450A sonicator with a cup horn for 30 seconds. Samples diluted (10 fold) in PBS and plated using a spiral systems autoplate 4000 spiral plater on Veillonella Agar.
Time Frame: 14 days
Measure: Log Mean (Standard Error); unit: log CFU (Colony forming units)
Arm/Group | Placebo | Active Comparator | Experimental
Number analyzed (Participants) | 24 | 24 | 24
log CFU (Colony forming units) | -0.0732 (0.0351) | 0.2579 (0.0426) | -0.0676 (0.0294)
Statistical Analysis 1: Comparison: Placebo vs Active Comparator vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Placebo - Fluoride Control: Fluoride only toothpaste (Crest Anti-Cavity)
- Active Comparator: Active Comparator toothpaste containing fluoride/triclosan/copolymer (Total)
- Experimental: Experimental test product (stannous fluoride toothpaste)
Arm/Group | Placebo - Fluoride Control | Active Comparator | Experimental
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less